CLINICAL TRIAL: NCT06452940
Title: Effects of Clinical Pilates Exercises on Glycemic Control, Blood Lipids and Physical Fitness Parameters in Individuals With Prediabetes: Controlled Study
Brief Title: Effects of Clinical Pilates Exercises on Glycemic Control, Blood Lipids and Physical Fitness Parameters in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKaraman
Record Dates: First submitted 2024-05-16; First posted 2024-06-11 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Prediabetic State
Keywords: Prediabetics; Exercise; Glycemic Control; Blood Glucose
MeSH Terms: conditions — Prediabetic State; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Diabetes education will be given at the beginning and ways to prevent type 2 diabetes will be explained.Evaluation will be made at the beginning and at the end of 16 weeks.
- Exercise Group (Experimental): Diabetes education will be given at the beginning and ways to prevent type 2 diabetes will be explained.Clinical pilates exercises will be performed.It will consist of a warm-up, main exercise and a cool-down period.Exercises will start with 10 repetitions and will be gradually increased in 3-week periods.Before the exercise training begins, all participants will be informed about clinical pilates and its basic principles will be explained. In the first session; The 5 key elements of pilates that should not be disrupted during exercises are; breathing, centering, rib cage placement, shoulder placement, head and neck placement will be taught. Exercise program will be done 3 days a week for 16 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A 16-week clinical pilates exercise program will be applied 3 days a week for 60 minutes each session. It will consist of a warm-up, main exercise and a cool-down period.Exercises will start with 10 repetitions and will be gradually increased in 3-week periods.
  Other Names: Clinical pilates
  Arms: Exercise Group

SUMMARY:
To examine the effects of clinical pilates exercise on glycemic control, blood lipids and physical fitness parameters in prediabetics. Subjects will be divided into two groups through randomization.Subjects in the 1st group will be included in the control group and will continue their routine. Subjects in the 2nd group will be given clinical pilates exercise training. All subjects will be evaluated at the start of treatment, and week 16.

DETAILED DESCRIPTION:
Prediabetes refers to the middle stage of dysglycemia in the process from normoglycemia to diabetes. It is diagnosed by laboratory measurement of fasting blood glucose, glycosylated hemoglobin or blood glucose 2 hours after loading.

The increasing prevalence of prediabetes worldwide is an important public health problem. However, active recognition and treatment of prediabetes has lagged because clinicians do not see it as a disease state that needs to be addressed. Low levels of physical activity and physical fitness (both cardiovascular and musculoskeletal) are significant, independent and modifiable risk factors for the development of type 2 diabetes, and lifestyle changes, including exercise training, now represent a central strategy in diabetes prevention.

Hypotheses:

H1: Clinical pilates training given to individuals with prediabetes has no effect on glycemic control.

H2: Clinical pilates training given to individuals with prediabetes has no effect on blood lipids.

H3: Clinical pilates training given to individuals with prediabetes has no effect on physical fitness parameters.

H4: Clinical pilates training given to individuals with prediabetes has no effect on exercise beliefs.

Material and Method:

The study will be conducted on subjects diagnosed with prediabetes by specialist physician.Subjects who meet the inclusion and exclusion criteria and sign the informed consent form will be randomly divided into two different groups by random allocation program.

According to the power analysis made using the G-Power program; Assuming that the nonparametric ANOVA test will be used for the comparison between the 2 groups, and a total of 42 people will be included in the calculation made by taking Cohen d=0.40, α=0.05, β=0.20, 21 in each group.

Subjects will be divided into two groups through randomization. Randomization will be done with random allocation software program. Both groups will be informed about ways to prevent diabetes. Subjects in group 1 will continue their routine for 16 weeks. Subjects in the 2nd group will be given clinical pilates exercise training. Exercise training will continue for 16 weeks. Clinical pilates exercises will be 3 days a week. All participants will be evaluated before treatment, and 16 weeks.

Evaluations to be applied to the Subject:

Socio-demographic Form: Age, gender, height, body weight, dominant side, marital status, educational status, occupation, diseases in the past and family history, alcohol and cigarette consumption, year of prediabetes diagnosis, medication use, and history of surgery will be questioned from the individuals who will participate in the study.

Body composition measurement:

With bioelectrical impedance analyzer; Weight, body fat percentage, total body water, fat mass, lean body mass will be measured. Additionally, waist and hip circumferences will be measured with a tape measure and the waist/hip ratio will be calculated.

Biochemical tests:

People's HbA1c, fasting glucose, fasting insulin, HOMA-IR, HDL, LDL, vitamin D, Triglyceride and total cholesterol values will be questioned based on blood analyzes performed during routine doctor's checks.

Muscle strength measurement:

Grip strength will be measured with a hand-grip dynamometer. The patient will be asked to sit with an upright back and grasp and squeeze the dynamometer with the dominant side hand. The best value will be recorded by repeating three times.

Muscle strength of the upper and lower extremity muscles will be measured using a digital hand-held dynamometer. In order to ensure that the movement is revealed correctly in the measurements, the individuals will be asked to perform submaximal contraction against the hand of the evaluator and the evaluation will be started after the test trial is performed. The best value will be recorded after three repetitions.

Evaluation of Functional Strength of Core Muscles:

Sit-ups and Modified Push-ups tests will be performed. Measurements will be made using a stopwatch and the number of repetitions performed by individuals within 30 seconds will be recorded.

Endurance Assessment A 30-second sit and stand test will be performed to assess lower extremity endurance. McGill protocol will be applied to assess core endurance. This protocol includes trunk flexion, lateral bridge, modified "Biering-sorensen", prone bridge tests.

30 Second Sit and Stand Test: The participant will be asked to sit on a chair with a backrest and cross their arms over their shoulders. Then he/she will be told to sit up and get up from the chair with our start command, keeping the time for 30 seconds. The number of sit-ups during this time will be recorded.

Trunk Flexion Test: The trunk will be flexed 60°, knees and hips will be flexed 90°. The arms will be crossed over the chest and the participants will be asked to maintain this position for as long as possible.

Lateral Bridge Test: It will be performed lying on the mat on the side. Participants will be asked to lift their hips upwards and maintain this position.

Modified "Biering-sorensen" Test: It will be performed in prone position on the treatment table. The pelvis, hips and knees will be fixed on the treatment table up to the level of the spina iliaca anterior superior. Participants will be asked to maintain the body position for as long as possible by crossing their arms across the chest.

Prone Bridge Test: Participants will be asked to lift their torso upwards by placing their weight on their forearms and toes in a prone, elbow flexion position. Tests will be terminated when positions are disrupted. Measurement results will be recorded in seconds.

Flexibility Assessment:

Sit-Reach Test and Lateral Flexion Test will be performed. Sit-Reach Test: In the test, a ruler will be placed on a cube with a side of 30 cm. The participant will be asked to rest the sole of his/her foot on the cube in a long sitting position and reach out on the ruler with both hands and knees in extension. The edge of the cube will be taken as 0 and values above it will be taken as positive and values below it will be taken as negative. The test will be repeated three times and the highest value will be recorded.

Lateral Flexion Test: While the participant stands with arms straight next to the trunk, the 3rd fingertip projection on both sides will be marked on the body. The participant will be asked to tilt the body to one side first and the projection of the 3rd fingertip will be marked and the distance between the first projection will be noted in cm. Measurements will be made on both sides.

Balance Assessment:

Fullerton advanced balance (FAB-T) scale will be used. The FAB-T is a scale designed to assess changes in different dimensions of balance. The performance-based FAB-T scale consists of 10 items assessing functional balance (static and dynamic) status. Each test is scored between 0-4, with a maximum score of 40 and a minimum score of 0. A higher score represents better balance.

Exercise Beliefs Assessment:

Exercise will be evaluated with the benefits/obstacles scale. The Turkish validity and reliability of the scale was conducted by Ortabağ et al. The scale, which has a Cronbach's alpha coefficient of 0.95, is a 4-point Likert-type scale and is answered from 4 (strongly agree) to 1 (strongly disagree). Consisting of 43 questions, the total score of the scale is between 43-172. It has two sub-dimensions as Exercise Benefit Scale and Exercise Barrier Scale. Each sub-dimension can be evaluated separately. The total score of the benefit scale is between 29-116 and the total score of the barrier scale is between 14-56. A high total score on the Exercise Benefit Scale indicates that the individual has a good perception of exercise benefit, while a high total score on the Exercise Barrier Scale indicates that the individual has a high perception of exercise barrier.

All assessments will be made before treatment, and week 16.

Interventions:

1. Group (Control): Subjects will continue their routine.
2. Group (Clinical Pilates Exercises): A 16-week clinical pilates exercise program will be applied 3 days a week for 60 minutes each session. It will consist of a warm-up, main exercise and a cool-down period.Before the exercise training begins, all participants will be informed about clinical pilates and its basic principles will be explained. In the first session; The 5 key elements of pilates that should not be disrupted during the exercises are; breathing, centering, rib cage placement, shoulder placement, head and neck placement will be taught. Exercises will start with 10 repetitions and will be gradually increased in 3-week periods.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Prediabetes
* Being between the ages of 30-60
* Not having received physiotherapy in the last 6 months
* Being physically inactive (<150 min/week or <600 MET/week according to the International Physical Activity Survey Short Version)

Exclusion Criteria:

* Having a history of type 2 diabetes
* Taking any supplements to maintain weight control
* Having a history of acute trauma affecting the movement system within the last month
* Presence of orthopedic/neurological/cardiopulmonary disease affecting the movement system
* Pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
The glycosylated hemoglobin A1c | at baseline and at the end of the 16th week
  An A1C test result reflects your average blood sugar level for the past two to three months. Specifically, the A1C test measures what percentage of hemoglobin proteins in your blood are coated with sugar (glycated). Hemoglobin proteins in red blood cells transport oxygen.
  The higher your A1C level is, the poorer your blood sugar control and the higher your risk of diabetes complications.

SECONDARY OUTCOMES:
Fasting Blood Glucose | at baseline and at the end of the 16th week
  The expected values for normal fasting blood glucose concentration are between 70 mg/dL (3.9 mmol/L) and 100 mg/dL (5.6 mmol/L). When fasting blood glucose is between 100 to 125 mg/dL (5.6 to 6.9 mmol/L) changes in lifestyle and monitoring glycemia are recommended.
Fasting insulin | at baseline and at the end of the 16th week
  Fasting insulin value will be checked based on blood analyses performed during routine doctor controls.
HOMA-IR | at baseline and at the end of the 16th week
  HOMA-IR value will be checked based on blood analyses performed during routine doctor controls.
HDL, LDL | at baseline and at the end of the 16th week
  values will be checked based on blood analyses performed during routine doctor controls.
Vitamin D | at baseline and at the end of the 16th week
  Vitamin D, value will be checked based on blood analyses performed during routine doctor controls.
Triglyceride | at baseline and at the end of the 16th week
  Triglyceride, value will be checked based on blood analyses performed during routine doctor controls.
Total cholesterol | at baseline and at the end of the 16th week
  Total cholesterol, value will be checked based on blood analyses performed during routine doctor controls.
Body composition measurement | at baseline and at the end of the 16th week
  Weight, body fat percentage, total body water, fat mass, fat mass, lean body mass will be measured with a bioelectrical impedance analyzer.
Waist-hip ratio | at baseline and at the end of the 16th week
  Waist and hip circumference will be measured with a tape measure and waist/hip ratio will be calculated.
Grip Strength | at baseline and at the end of the 16th week
  Grip strength will be measured with a hand-grip dynamometer. The patient will be asked to sit with his/her back straight and grasp and squeeze the dynamometer with the dominant side hand. The best value will be recorded by repeating three times
Muscle Strength | at baseline and at the end of the 16th week
  Muscle strength of the upper and lower extremity muscles will be measured using a digital hand-held dynamometer. In order to ensure that the movement is correctly revealed in the measurements, the individuals will be asked to perform submaximal contraction against the evaluator's hand and the evaluation will be started after the test trial is performed. The best value will be recorded after three repetitions
Functional Strength of Core Muscles | at baseline and at the end of the 16th week
  Sit-ups and modified push-up tests will be performed. Measurements will be made using a stopwatch and the number of repetitions performed by individuals within 30 seconds will be recorded
Sit-up Test | at baseline and at the end of the 16th week
  Sit-up tests will be performed for the functional strength of core muscles. Measurements will be made using a stopwatch and the number of repetitions performed by individuals within 30 seconds will be recorded
Modified push-up Test | at baseline and at the end of the 16th week
  Modified push-up tests will be performed for functional strength of core muscles. Measurements will be made using a stopwatch and the number of repetitions performed by individuals within 30 seconds will be recorded
Lower Extremity Endurance | at baseline and at the end of the 16th week
  A 30-second sit and stand test will be performed to assess lower extremity endurance.
  McGill protocol will be applied to evaluate core endurance. This protocol includes trunk flexion, lateral bridge, modified "Biering-sorensen", prone bridge tests.Tests will be terminated when the positions are disturbed. The measurement results will be recorded in seconds.
Core Endurance | at baseline and at the end of the 16th week
  McGill protocol will be applied to evaluate core endurance. This protocol includes trunk flexion, lateral bridge, modified "Biering-sorensen", prone bridge tests.Tests will be terminated when the positions are disturbed. The measurement results will be recorded in seconds.
Sit-Reach Test | at baseline and at the end of the 16th week
  SRT will be performed for flexibility. The test will be repeated three times and the highest value will be recorded.
Lateral Flexion Test | at baseline and at the end of the 16th week
  LFT will be performed for flexibility.The test will be repeated three times and the highest value will be recorded.
Balance | at baseline and at the end of the 16th week
  The Fullerton advanced balance (FAB-T) scale will be used.
Exercise Beliefs | at baseline and at the end of the 16th week
  Exercise beliefs will be assessed with the exercise benefits/barriers scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşen Karaman, MSc, Principal Investigator — EMU; Ender Angın, PhD, Study Director — EMU
Locations (1):
- Eastern Mediterranean University, Mersin, Famagusta, Turkey (Türkiye)

REFERENCES:
- [Background] ADA(Am.DiabetesAssoc.).2020.2.Classificationanddiagnosisofdiabetes:StandardsofMedicalCare in Diabetes-2020. Diabetes Care 43(Suppl. 1):S14-31
- [Background] Echouffo-Tcheugui JB, Selvin E. Prediabetes and What It Means: The Epidemiological Evidence. Annu Rev Public Health. 2021 Apr 1;42:59-77. doi: 10.1146/annurev-publhealth-090419-102644. Epub 2021 Dec 23. PMID 33355476